CLINICAL TRIAL: NCT03929289
Title: The Visuo-attentional Mediator of Social Facilitation
Acronym: VAMOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL19_0268; 2019-A01027-50 (Other: ID-RCB)
Record Dates: First submitted 2019-04-12; First posted 2019-04-26 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Social Facilitation
Keywords: Functional Magnetic Resonance Imaging (fMRI); Healthy Subjects
MeSH Terms: conditions — Social Facilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Social Facilitation (Experimental): Cognitive tasks during the 2 functional Magnetic Resonance Imaging (fMRI) observed or not by a subject's known peer.
  Interventions: Behavioral: Social Facilitation

INTERVENTIONS:
Behavioral: Social Facilitation — During the functional Magnetic Resonance Imaging (fMRI) scans, the subject will perform cognitive tasks measuring eye movements and attention alternatively observed by a familiar peer (in an adjacent room) or not.

SUMMARY:
Social psychology has long established that the mere presence of others influences the investigator's individual behavior and performance. "Social facilitation" refers to any improvement or deterioration of performance due to the presence of others. For more than a century, social psychology has acquired a solid knowledge of the principles governing this fundamental form of social influence.

But the underlying mechanism of social facilitation remains debated, as behavior alone cannot identify it with certainty. This major unresolved problem makes it particularly difficult to translate laboratory results on social facilitation into real applications in areas such as school or work, where others are ubiquitous. The purpose of this study will therefore be to identify the mediator of social facilitation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18 to 35 years old
* Signed written informed consent
* Insurance coverage

Exclusion Criteria:

* Neurological or psychiatric or ophthalmological disorder
* Non-stabilized medical condition
* Ongoing treatment with drugs that affect the central nervous system

  * Uncorrected visual inadequacy
  * No fluency in French reading
  * Pregnant and / or breastfeeding woman, this exclusion criterion will be sought by questioning the subject
  * Subject commonly in care in a health or social facility for purposes other than that of research
  * Subject under guardianship
  * Subject deprived of liberty by a judicial or administrative decision
  * Incompatibility with the Magnetic Resonance Imaging (MRI) examination determined by answering the following questions:
* Carrier of a neurological stimulator, cardiac (battery) or defibrillator
* Carrier of a cardiac prosthesis (valve, stent ...) or vascular
* Holder of intracranial clips or clamps (staples)
* Carrier of a cerebrospinal fluid bypass
* Presence of metal chips in the eyes
* Metal prosthesis carrier (teeth, knees)
* Pump carrier or infusion system
* Presence of metal tattoo near the head
* Presence of permanent makeup
* Claustrophobia or respiratory disorders

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Brain activation | 50 minutes
  Cerebral Blood Oxygenation Level-Dependent (BOLD) signals

SECONDARY OUTCOMES:
Behavioral performances | 50 minutes
  pupillary diameter
Behavioral performances | 50 minutes
  error rate
Behavioral performances | 50 minutes
  reaction time
Behavioral performances | 50 minutes
  oculomotor kinematic parameters: velocity of saccades.
Behavioral performances | 50 minutes
  oculomotor kinematic parameters: duration of saccades.
Behavioral performances | 50 minutes
  oculomotor kinematic parameters: precision of saccades.

CONTACTS AND LOCATIONS:
Overall Officials: Denis PELISSON, Principal Investigator — Centre de Recherche en Neuroscience de Lyon
Locations (1):
- Centre de Recherche en Neuroscience de Lyon, Bron, France

REFERENCES:
- [Background] Tricoche L, Royer d'Halluin M, Meunier M, Pelisson D. Neural bases of social facilitation and inhibition: how peer presence affects elementary eye movements. Soc Cogn Affect Neurosci. 2025 Jun 17;20(1):nsae079. doi: 10.1093/scan/nsae079. PMID 39506559